CLINICAL TRIAL: NCT05510258
Title: Comparison of Routine Physical Therapy With and Without Core-stability Exercises on Dynamic Sitting Balance and Trunk Control in Sub-acute Ischemic Stroke Patient
Brief Title: Comparison of Routine and Core-stability Exercises on Dynamic Sitting Balance and Trunk Control in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-UOL-FAHS/718-XV/2020
Record Dates: First submitted 2022-08-15; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Ischemic Stroke, Acute
MeSH Terms: conditions — Ischemic Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Two groups control and experimental included
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): core-stability exercises therapy given with conventional therapy
  Interventions: Other: Physiotherapy
- control group (Other): only conventional therapy given
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — TWO GROUPS CONTROL ND EXPERIMENTAL

SUMMARY:
This is ROM trail study. Data collected from Rabbani Hospital Lahore . in this study total two groups included control and experimental and sample size was 48 and 24 persons divided in each groups as well. Informed consent was taken from the recruited subjects. Two scales BBS and TIS used to measure the outcomes. Data analyse by ssps V21.0 with a significant level of p valued 0.05. Results were in the favour of experimental group.

DETAILED DESCRIPTION:
This is ROM trail study. Data collected from Physiotherapy department of Rabbani Hospital Lahore . In this study total two groups included control and experimental and sample size was 48 and 24 persons randomly allocated in each groups as well. In control group conventional therapy given while in experimental group core-stability exercises with conventional therapy given to the patients. while the duration of therapy was 45 minutes per day for 8 weeks. Informed consent was taken from the recruited subjects. Two scales BBS and TIS used to measure the outcomes. Only having first episode of sub-acute stoke patients and diagnosed by Neuro-physician were included in study. Data entered and analysed by SSPS V21.0 with a significant level of p valued 0.05. and the results were in the favour of study means experimental group.

ELIGIBILITY:
* Inclusion Criteria:

  * Sub-Acute ischemic and stroke diagnosed by neuro-physican having 1st episode
  * Patients in sub-acute stage (2-12 weeks)
  * Patients who can follow the instruction according to mini mental scale < 7
  * Minimum score of a patient on burg balance and trunk impairment scale to enter in rehab unit and include in any research i-e TIS < 2 in scoring and BBS < 4 minimum scoring.
* Exclusion Criteria:

  * Recurrent stroke
  * Subjects with radiating pain or nerve root involvement
  * Diagnosed by any neurological condition other than stroke, or other clinical comorbidity that affect the trunk balance.
  * Patient unable to follow the instructions
  * Comprehension deficits that prevented them from following verbal commands
  * Unconscious patient

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Berg balance scale at week 4 | Baseline and 4 weeks
  Berg balance scale(BBS) used clinical test of a person's static and dynamic balance abilities. BBS comprises a set of 14 items which includes unsupported sitting to unsupported standing and weight shifting while standing unsupported.
  * Lower score =1 (Sitting to standing)
  * Higher score=14 (weight shifting while standing)
Change from baseline in Trunk impairment scale at week 4 | Baseline and 4 weeks
  The Trunk Impairment Scale (TIS) is a tool to measure motor impairment of the trunk after stroke. TIS scores on a range from 0 to 23. Static sitting balance, Dynamic sitting balance and Co-ordination will be evaluated by this scale.
  * Static sitting balance=7
  * Dynamic sitting balance=10
  * Co-ordination=6

CONTACTS AND LOCATIONS:
Overall Officials: Rabbani Hospital, Study Chair — PMDC
Locations (1):
- Duaa Awais, Lahore, Punjab Province, Pakistan